CLINICAL TRIAL: NCT03931772
Title: Pilot Study Evaluating the Feasibility and Effects of an Innovative Automated Hypnosis Intervention for Smoking Cessation and Pain and Stress Reduction
Brief Title: Online Automated Self-Hypnosis Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Spiegel, Jack, Lulu and Sam Willson Professor and Associate Chair of Psychiatry & Behavioral Sciences, Director Center on Stress and Health, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 42124
Record Dates: First submitted 2019-04-02; First posted 2019-04-30 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Smoking; Pain; Stress
MeSH Terms: conditions — Smoking; Pain

STUDY DESIGN:
Intervention Model Description: This is a pilot, open trial evaluating a novel automated hypnosis intervention for smoking cessation and pain and reduction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Automated Self-Hypnosis Intervention for Smoking Cessation (Experimental): Participants will first try this intervention at their Baseline visit following an assessment of trait hypnotizability. After being guided through the program by their experimenter (i.e., set-up procedures in addition to the actual hypnotic exercise) participants will provide initial feedback on the program through a series of questions. The entire appointment will take approximately one hour and will take place at The Center on Stress and Health. Participants will be provided with the Amazon Alexa device to take home (necessary for using the program), or the interactive Reveri (www.reveri.com) mobile app. After the lab visit participants will continue using the intervention at home as needed throughout the 24 months of study participation (recommended every few hours or whenever they feel the urge to smoke). Furthermore, participants will be taking an online 15-minute survey at the baseline visit, and then 1, 3, 6, 12 and 24-month online follow-up surveys at home.
  Interventions: Behavioral: Automated Self-Hypnosis
- Automated Self-Hypnosis Intervention for Pain Reduction (Experimental): Participants will first try this intervention at their Baseline visit following an assessment of trait hypnotizability. After being guided through the program by their experimenter (i.e., set-up procedures in addition to the actual hypnotic exercise) participants will provide initial feedback on the program through a series of questions. The entire appointment will take approximately one hour and will take place at The Center on Stress and Health, or remotely during the COVID-19 pandemic. Participants will be provided with the Amazon Alexa device to take home (necessary for using the program), or the interactive Reveri (www.reveri.com) mobile app. After the lab or remote visit participants will continue using the intervention at home as needed (recommended every few hours or whenever they experience an increase in pain). Furthermore, participants will be taking an online 15-minute survey at the baseline visit, and then 1, 3, 6, 12 and 24-month online follow-up surveys at home.
  Interventions: Behavioral: Automated Self-Hypnosis
- Automated Self-Hypnosis Intervention for Stress Reduction (Experimental): Participants will first try this intervention at their Baseline visit following an assessment of trait hypnotizability. After being guided through the program by their experimenter (i.e., set-up procedures in addition to the actual hypnotic exercise) participants will provide initial feedback on the program through a series of questions. The entire appointment will take approximately one hour and will take place at The Center on Stress and Health, or remotely during the COVID-19 pandemic. Participants will be provided with the Amazon Alexa device to take home (necessary for using the program), or the interactive Reveri (www.reveri.com) mobile app. After the lab or remote visit participants will continue using the intervention at home as needed (recommended every few hours or whenever they experience an increase in stress). Furthermore, participants will be taking an online 15-minute survey at the baseline visit, and then 1, 3, 6, 12 and 24-month online follow-up surveys at home.
  Interventions: Behavioral: Automated Self-Hypnosis

INTERVENTIONS:
Behavioral: Automated Self-Hypnosis — Self-Hypnosis will be delivered through an interactive application administered through Amazon Alexa or Reveri.com.

SUMMARY:
After developing professional quality materials (audio) for an affordable automated self-hypnosis intervention program for facilitating smoking cessation, stress and pain reduction, researchers aim to gain qualitative reviews of this program, and test its initial feasibility and effects on smoking cessation and reduction in pain and stress.

In addition, this study seeks to determine whether higher hypnotizability, as measured by the Hypnotic Induction Profile (assessed at baseline), is a moderator of improved outcome in these conditions.

DETAILED DESCRIPTION:
The investigators are interested in recruiting individuals who report that they smoke cigarettes daily and are motivated to make a serious attempt at quitting, and individuals who report experiencing pain or stress, who are willing to try to use the hypnosis intervention and provide feedback regarding their experience with the intervention.

The original intervention is an interactive hypnosis tool, developed by Reveri Health, utilizing periodic questions and answers to personalize the session progression and emulate the conversational nature of an in-person session designed based upon decades of clinical hypnosis research and experience at the Stanford Center on Stress and Health. The intervention is delivered through the Amazon Alexa platform's beta testing tool. Participants will be provided with the Alexa Dot device, which is sold by Amazon and widely used by consumers. Later on, research participants will have the option of using an Alexa-supported smartphone device without the Alexa Dot speaker. Those enrolled later in the study will instead be offered the use of the interactive app also developed by Reveri (www.reveri.com) independent of the Alexa platform. What will be specific to this pilot is the hypnosis training approach, including the interactive nature of the program. The structure and the content of the hypnosis training program will be the same across the 3 mentioned modes of administration. The user interface for the app is the main difference.

ELIGIBILITY:
Inclusion/Exclusion criteria for the three arms, with exceptions noted below:

Inclusion Criteria:

* 18 years or older
* Able to read and understand English
* For the smokers, desire to quit smoking (specifically, report a motivation of ≥ 5 out of 10 to quit smoking on a 10-point Likert-type scale), and report being a daily smoker for at least one year, smoking an average ≥ 5 cigarettes per day
* For the pain group, report suffering from chronic pain syndromes, such as fibromyalgia or chronic low back pain
* For the stress group, report experiencing moderate to extreme stress or anxiety in the past month
* Having access to wireless internet connection or mobile data

Exclusion Criteria:

* Meeting criteria for drug abuse, including use of dissociative anesthetics, hallucinogens, opioids, cocaine, or amphetamine within the last 3 months
* Severe psychiatric or structural brain disease (i.e. psychosis, stroke with functional impairment, dementia) or current/recent risk to self
* Hearing impairment that would impede ability to listen the auditory intervention
* Major illnesses impacting the study results
* For smokers, currently taking Wellbutrin, Chantix, or other pharmacological smoking cessation aids that could confound results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Rate of Self-reported smoking cessation | Baseline through month 24
  The question, with a dichotomous (yes/no) response, "Have you succeeded in stopping smoking completely?" will be asked via online survey. Researchers will use responses of "Yes" to indicate abstinence.
Change in Brief Pain Inventory-Pain Interference Score | Baseline through month 24
  Participant-reported outcome. Scores range from 0-10 and higher scores indicate worst pain.
Change in Brief Pain Inventory-Pain Severity Score | Baseline through month 24
  Participant-reported outcome. Scores range from 0-10 and higher scores indicate worst pain.
Change in McGill Pain Questionnaire | Baseline through month 24
  Participant-reported outcome. Scores range from 0-78 and the higher the pain score the greater the pain.
Change in PROMIS SF v1.0 Pain Interference 4a short form | Baseline through month 24
  Participant-reported raw scores are converted to T-scores where T = 50 is the population mean and T = 40 and 60 are 1 SD below and above the population mean respectively. Higher T scores indicate higher pain.
Change in PROMIS Global Pain Intensity (Pain Intensity 1a) | Baseline through month 24
  Participant-reported outcome. Scores range from 0 (no pain) to 10 (Worst imaginable pain).
Change in Perceived Stress Scale | Baseline through month 24
  Participant-reported outcome. Scores range from 10-50; higher scores indicate higher stress.
Change in Stanford Acute Stress Reaction Questionnaire | Baseline through month 24
  Participant-reported outcome. Scores range from 0 to 150 with higher scores indicating higher acute stress.
Change in Impact of Event Scale - Revised | Baseline through month 24
  Participant-reported outcome evaluating subjective stress caused by traumatic events, where scores range from 0-88 and higher scores indicate higher subjective stress.
Change in Positive and Negative Affect Scale-Negative Affect Scale Score | Baseline through month 24
  Participant-reported outcome. This reporting tool has positive and negative affect scales; the negative affect scale is a primary outcome measure in this study. Scores range from 10-50 and higher scores indicate higher negative affect.
Change in State-Trait Anxiety Inventory Form X | Baseline through month 24
  Participant-reported outcome. Scores range from 20-80 and higher scores indicate higher state anxiety.
Change in State-Trait Anxiety Inventory Form Y | Baseline through month 24
  Participant-reported outcome. Scores range from 20-80 and higher scores indicate higher trait anxiety.

SECONDARY OUTCOMES:
Rate of smoking reduction over time | Baseline through month 24
  Change in the number of self-reported daily cigarettes smoked at follow-ups will be examined.
Change in PROMIS SF v1.0 Physical Function 4a short form | Baseline through month 24
  Participant-reported raw scores are converted to T-scores where T = 50 is the population mean and T = 40 and 60 are 1 SD below and above the population mean respectively. Higher T scores indicate higher physical function.
Change in PROMIS SF v1.0 Anxiety 4a short form | Baseline through month 24
  Participant-reported raw scores are converted to T-scores where T = 50 is the population mean and T = 40 and 60 are 1 SD below and above the population mean respectively. Higher T scores indicate higher anxiety.
Change in PROMIS SF v1.0 Depression 4a short form | Baseline through month 24
  Participant-reported raw scores are converted to T-scores where T = 50 is the population mean and T = 40 and 60 are 1 SD below and above the population mean respectively. Higher T scores indicate higher depression.
Change in PROMIS SF v1.0 Fatigue 4a short form | Baseline through month 24
  Participant-reported raw scores are converted to T-scores where T = 50 is the population mean and T = 40 and 60 are 1 SD below and above the population mean respectively. Higher T scores indicate higher fatigue.
Change in PROMIS SF v1.0 Sleep Disturbance 4a short form | Baseline through month 24
  Participant-reported raw scores are converted to T-scores where T = 50 is the population mean and T = 40 and 60 are 1 SD below and above the population mean respectively. Higher T scores indicate higher sleep disturbance.
Change in PROMIS SF v1.0 Ability to Participate in Social Roles and Activities 4a short form | Baseline through month 24
  Participant-reported raw scores are converted to T-scores where T = 50 is the population mean and T = 40 and 60 are 1 SD below and above the population mean respectively. Higher T scores indicate higher ability to participate in social roles and activities.
Change in Positive and Negative Affect Scale-Positive Affect Scale Score | Baseline through month 24
  Participant-reported outcome. This reporting tool has positive and negative affect scales; the positive affect scale is a secondary outcome measure in this study. Scores range from 10-50 and higher scores indicate higher positive affect.
Change in Brief Cope Scale | Baseline through month 24
  Participant-reported outcome. Scores range from 2-8 and higher scores indicate greater ability to cope.
Change in Pittsburgh Sleep Quality Index | Baseline through month 24
  Participant-reported outcome of change in sleep quality. Scores range from 0-21 and higher scores indicate worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford Medicine - Psychiatry and Behavioral Sciences, Palo Alto, California
  - Dept. of Psychiatry, Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No